CLINICAL TRIAL: NCT03834220
Title: A Phase II Basket Study of the Oral Selective Pan-FGFR Inhibitor Debio 1347 in Subjects With Solid Tumors Harboring a Fusion of FGFR1, FGFR2 or FGFR3
Brief Title: Basket Trial in Solid Tumors Harboring a Fusion of FGFR1, FGFR2 or FGFR3- (FUZE Clinical Trial)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lower antitumor activity than expected
Sponsor: Debiopharm International SA (Industry)
Collaborators: Caris Life Sciences (Industry); Optimal Research (Just In Time sites) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1347-201; 2018-003584-53 (EudraCT Number)
Record Dates: First submitted 2019-02-04; First posted 2019-02-07 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — CH5183284

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Debio 1347 (Biliary Tract Cancer) (Experimental): Participants with biliary tract cancer were included in this cohort to receive Debio 1347 80 milligrams (mg) tablets, orally, once daily (QD), from Day 1 to Day 28 in 28-day cycles until the occurrence of disease progression or unacceptable toxicity (up to a median duration of 20 weeks).
  Interventions: Drug: Debio 1347
- Cohort 2: Debio 1347 (Urothelial Cancer) (Experimental): Participants with urothelial cancer were included in this cohort to receive Debio 1347 80 mg tablets, orally, QD, from Day 1 to Day 28 in 28-day cycles until the occurrence of disease progression or unacceptable toxicity (up to a median duration of 5.86 weeks).
  Interventions: Drug: Debio 1347
- Cohort 3: Debio 1347 (All Other Solid Tumor Histologies) (Experimental): Participants with all other solid tumor histologies were included in this cohort to receive Debio 1347 80 mg tablets, orally, QD, from Day 1 to Day 28 in 28-day cycles until the occurrence of disease progression or unacceptable toxicity (up to a median duration of 8.14 weeks).
  Interventions: Drug: Debio 1347

INTERVENTIONS:
Drug: Debio 1347 — Debio 1347 oral tablets.

SUMMARY:
The primary objective of this study is to assess the efficacy of Debio 1347 in terms of objective response rate (ORR) in participants with solid tumors harboring fibroblast growth factor receptor (FGFR)1-3 gene fusion/rearrangement.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed advanced solid tumor
* Radiographic progression on prior systemic therapy; prior localized therapy (i.e., radiation, ablation, embolization) is allowed provided radiographic progression out-of-field or in the treatment, field is shown
* Locally-advanced (unresectable) or metastatic disease harboring an FGFR1-3 gene fusion/rearrangement potentially leading to a functional FGFR aberrant protein, identified through local and/or central molecular assay

Exclusion Criteria:

* History of hypersensitivity to any of the excipients in the Debio 1347 formulation
* History and/or current evidence of ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, myocardia, or lung, excepting calcified lymph nodes, lung nodules and asymptomatic vascular or cartilage/tendon calcifications
* Administration of any investigational agent within 2 weeks prior to initial dosing with Debio 1347 (3 weeks for immune checkpoint inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (105):
- United States (25):
  - Ironwood Cancer & Research Centers - Scottsdale, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Moores UCSD Cancer Center, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Sarcoma Oncology Center, Santa Monica, California
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Tulane University Cancer Center, New Orleans, Louisiana
  - The John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, Middletown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, Harrison, New York
  - Memorial Sloan-Kettering Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - UC Health, LLC., Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center - James Cancer Hospital, Columbus, Ohio
  - CTCA Cancer Treatment Centers, Tulsa, Oklahoma
  - West Penn - Allegheny Oncology Network, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - Fred Hutchinson/Seattle Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (4):
  - Southern Highlands Private Hospital, Bowral
  - Peninsula and Southeast Oncology (PASO), Frankston
  - Linear Clinical Research, B Block Sir Charles Gairdner Hospital, Nedlands
  - John Flynn Private Hospital, Tugun
- Austria (2):
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Brazil (4):
  - Hospital de Caridade de Ijuí, Avenida David J Martins, Ijuí
  - Hospital de Clínicas de Porto Alegre, Rio Grande
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, Avenida Doutor Arnaldo, São Paulo
- Bulgaria (3):
  - MHAT - Dobrich, Dobrich
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - MHAT "Serdika", EOOD, Sofia
- Croatia (2):
  - General Hospital Varazdin, Varaždin
  - University Hospital Centre, Sestre Milosrdnice, Zagreb
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Thomayerova nemocnice, Prague
- Denmark (3):
  - Ålborg Universitets Hospital, Aalborg
  - Herlev Hospital, Herlev
  - Odense Universitetshospital, Odense
- Finland (2):
  - Docrates Syöpäsairaala, Helsinki
  - Helsinki University Hospital, Helsinki
- France (6):
  - ICO - Site Paul Papin, Angers
  - CHU Bordeaux - Hôpital Saint André, Groupe Hospitalier Sud - Hôpital Haut-Lévêque, Bordeaux
  - Centre Oscar Lambret, Lille
  - Groupe Hospitalier Sud - Hôpital Haut Lévêque, Pessac
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Greece (4):
  - General Hospital of Athens Laiko, Athens
  - General Hospital of Athens of Chest Diseases "SOTIRIA", Athens
  - General Hospital of Athens "Alexandra", Athens
  - University General Hospital of Ioannina, Ioannina
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - Haga Ziekenhuis, The Hague
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Radiumhospitalet, Montebello, Oslo
- Philippines (3):
  - Cebu Doctors' University Hospital (CDUH), Research Office, Cebu City
  - Philippine General Hospital, Clinical Trial Unit Room 5, Medical Research Laboratory, Ermita
  - St. Luke's Medical Center, Human Cancer Biobank Research Center, Quezon City
- Poland (3):
  - Szpital Kliniczny im.Heliodora Swiecickiego Uniwersytetu Medycznego im.K. Marcinkowskiego w Poznaniu, Poznan
  - MTZ Clinical Research, Warsaw
  - Centrum Onkologii-Instytut im.M.Sklodowskiej Curie, Warsaw
- Romania (4):
  - S.C Delta Health Care S.R.L, Bucharest
  - S.C Medisprof S.R.L., Cluj-Napoca
  - S.C Centrul de Oncologie Sf. Nectarie S.R.L., Craiova
  - S.C Oncocenter Oncologie Clinica S.R.L., Timișoara
- Russia (6):
  - SBIH of Arkhangelsk region "Arkhangelsk Clinical Oncological Dispensary", Arkhangelsk
  - TSBHI "Altai Territorial oncological dispensary", Barnaul
  - LLC Evimed, Chelyabinsk
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - Tomsk Research Instutite of Oncology, Tomsk
- Singapore (2):
  - Singapore National Cancer Center (SNCC), Singapore
  - Tan Tock Seng Hospital, Communicable Disease Centre, Singapore
- South Korea (6):
  - Seoul National University Bundang Hospital, Department of Oncology Medical office, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, CRC Room, 3F, Gyeonggi-do
  - Gachon University Gil Medical Center, CRC Room, 18F, Artificial intelligence hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital (SNUH), Seoul
  - Ajou University Hospital, CRC room, Clinical Trial Center, Suwon
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (7):
  - Shuang Ho Hospital, New Taipei City
  - Taichung Veterans General Hospital, The Radiation Oncology Department, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital (TMUH), Taipei
  - Taipei Veterans General Hospital, Medical Science & Technology Building, Taipei
  - Linkou Chang-Gung Memorial Hospital, Taoyuan District
- Ukraine (3):
  - CI Dnipropetrovsk CMCH #4 of Dnipropetrovsk RC Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipro
  - SI V.T. Zaycev Institute of general & urgent surgery of National academy medical sciences of Ukraine, Department of purulent surgery, Kharkiv
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv
- United Kingdom (4):
  - Ninewells Hospital, Dundee
  - Guy's Hospital, London
  - Hammersmith Hospital, London
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 participants were enrolled at 31 investigational sites in the United States, France, Spain, Finland, Korea, Singapore, Australia, Bulgaria, Denmark, Norway, Russian Federation, Taiwan, and the United Kingdom from 22 March 2019 to 04 January 2022.
Pre-assignment Details: A total of 63 participants with solid tumors harboring FGFR1-3 gene fusion/rearrangement were enrolled into one of the 3 cohorts: Cohort 1: Biliary Tract Cancer (N=30), Cohort 2: Urothelial Cancer (N=4), Cohort 3: All Other Solid Tumor Histologies (N=29) to receive Debio 1347.
Period: Overall Study
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Started | 30 | 4 | 29
Completed | 0 | 0 | 0
Not Completed | 30 | 4 | 29
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 8 | 1 | 17
Not completed — Reason not Specified | 9 | 0 | 6
Not completed — Sponsor/EthicsCommittee Decided to Terminate Study | 10 | 1 | 4
Not completed — Withdrawal of Consent | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population consisted of all participants who received study drug.
Groups:
- Cohort 1: Debio 1347 (Biliary Tract Cancer): Participants with biliary tract cancer were included in this cohort to receive Debio 1347 80 mg tablets, orally, QD, from Day 1 to Day 28 in 28-day cycles until the occurrence of disease progression or unacceptable toxicity (up to a median duration of 20 weeks).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies) | Total
Number analyzed (Participants) | 30 | 4 | 29 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (12.21) | 55.3 (15.22) | 60.0 (12.58) | 59.3 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 2 | 16 | 34
  Male | 14 | 2 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 29 | 4 | 28 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 3 | 22 | 45
  Black or African American | 5 | 0 | 0 | 5
  Asian | 3 | 1 | 2 | 6
  Not Willing to Provide | 1 | 0 | 3 | 4
  Other | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Centrally Measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Criteria
Description: ORR was defined as the percentage of participants with a best overall response (BOR) of partial or complete response (PR or CR). BOR was defined as the best confirmed response observed from first administration of study drug until disease progression. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to disease progression or end of study (up to 1 year and 9 months)
Population: ITT Population consisted of all participants who received study drug. Overall number of participants analyzed is the number of participants with measurable disease and tumor assessment at Baseline.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1: Debio 1347 (Biliary Tract Cancer): Participants with biliary tract cancer were included in this cohort to receive Debio 1347 80 mg tablets, QD, from Day 1 to Day 28 in 28-day cycles until the occurrence of disease progression or unacceptable toxicity (up to a median duration of 20 weeks).
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 30 | 3 | 25
percentage of participants | 6.7 [1.2 to 19.5] | 0 [0.0 to 63.2] | 4.0 [0.2 to 17.6]

2. Secondary Outcome: Duration of Response (DOR) as Centrally Measured by Independent Review Committee (IRC)
Description: DOR was defined as the time from the date of the initial PR or CR to date of the first documented progression or death due to any cause. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to disease progression or end of study (up to 2 years and 9 months)
Population: ITT Population consisted of all participants who received study drug. Only participants with best overall response of CR or PR were analyzed for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 0 | 0 | 1
months |  |  | 5.55 [NA to NA] — The lower and upper limit of 95% confidence interval (CI) were not estimable due to insufficient number of participants with event.

3. Secondary Outcome: Disease Control Rate (DCR) as Centrally Measured by Independent Review Committee (IRC)
Description: DCR was defined as the percentage of participants with a BOR of confirmed CR, confirmed PR or stable disease (SD) ≥6 weeks. BOR was defined as the best confirmed response observed from first administration of study drug until disease progression. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD was defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Up to disease progression or end of study (up to 2 years and 9 months)
Population: ITT population consisted of all participants who received study drug. Percentages are rounded off to the nearest single decimal point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 30 | 4 | 29
percentage of participants | 63.3 [43.9 to 80.1] | 0 [0 to 60.2] | 34.5 [17.9 to 54.3]

4. Secondary Outcome: Progression-Free Survival (PFS) as Centrally Measured by Independent Review Committee (IRC)
Description: PFS was defined as the time from the start date of treatment to date of the first documented progression or death due to any cause.
Time Frame: From the start of the study up to disease progression or death (up to 2 years and 9 months)
Population: ITT population consisted of all participants who received study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 30 | 4 | 29
months | 3.68 [3.55 to 10.58] | 1.77 [0.95 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with event. | 1.84 [1.71 to 3.52]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start date of treatment to date of death due to any cause. Participants with no documented death were censored at the last date known to be alive.
Time Frame: Until death or loss to follow-up or end of study (up to 2 years and 9 months)
Population: ITT population consisted of all participants who received study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 30 | 4 | 29
months | NA [NA to NA] — The median, lower and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median, lower and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | 7.13 [4.30 to 11.37]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Assessed by National Cancer Institute Common Terminology Criteria (NCI CTCAE) v5.0 and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. A TEAE is defined as an AE that either starts or worsens in severity on or after the first administration of the study drug and within 30 days of the last administration of the study drug. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From first dose of study drug up to 30 days post last dose (Up to 2 years and 9 months)
Population: Safety Population consisted of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Debio 1347 (Biliary Tract Cancer): Participants with biliary tract cancer were included in this cohort to receive Debio 1347 80 mg tablets, orally, once daily QD, from Day 1 to Day 28 in 28-day cycles until the occurrence of disease progression or unacceptable toxicity (up to a median duration of 20 weeks).
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 30 | 4 | 29
Participants
  TEAEs | 30 | 4 | 28
  Serious TEAEs | 14 | 2 | 7

7. Secondary Outcome: Trough Concentration at Steady State (Ctrough,ss) of Debio 1347 in Plasma
Description: Geometric mean and geometric percent CV summary was estimated based on log-linear model.
Time Frame: Predose and post dose up to Cycle 2 Day 28 (each cycle length = 28 days)
Population: Pharmacokinetic (PK) Population included participants who received one or more doses of Debio 1347 and have at least one PK concentration result available. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 30 | 3 | 26
nanogram per millilitre (ng/mL) | 619.6 (100.0) | 306.8 (43.4) | 463.2 (127.3)

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Over the Dosing Interval at Steady State (AUCtau,ss) of Debio 1347 in Plasma
Description: Geometric mean and geometric percent CV summary was estimated based on log-linear model.
Time Frame: Predose and post dose up to Cycle 2 Day 28 (each cycle length = 28 days)
Population: PK Population included participants who received one or more doses of Debio 1347 and have at least one PK concentration result available. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram (h*ng)/mL
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 30 | 3 | 26
hour*nanogram (h*ng)/mL | 23326.7 (70.4) | 13999.0 (39.1) | 18192.1 (86.2)

9. Secondary Outcome: Correlation of Debio 1347 Plasma Concentration (C) and QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF)
Time Frame: Pre-dose on Days 14 and 28, and 1, 3, 7 hours post-dose on Day 28 of Cycle 1; pre-dose on Days 14 and 28, and 3 hours post-dose on Day 28 of Cycle 2 (each cycle length = 28 days)
Population: The study was terminated by sponsor and thus the analysis for this outcome measure was not deemed necessary and no data was collected.
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days post last dose (up to 2 years and 9 months)
Description: Safety Population consisted of all participants who received study drug. The all-cause mortality is reported for all participants enrolled in the study and who completed the study visits.
Arm/Group | Cohort 1: Debio 1347 (Biliary Tract Cancer) | Cohort 2: Debio 1347 (Urothelial Cancer) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies)
All-Cause Mortality (participants affected / at risk) | 9/30 | 1/4 | 17/29
Serious Adverse Events (participants affected / at risk) | 14/30 | 2/4 | 7/29
Other Adverse Events (participants affected / at risk) | 30/30 | 4/4 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Debio 1347 (Biliary Tract Cancer) (N=30) | Cohort 2: Debio 1347 (Urothelial Cancer) (N=4) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies) (N=29)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Biliary sepsis (Infections and infestations) | 2 | 0 | 0
Biliary tract infection (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Debio 1347 (Biliary Tract Cancer) (N=30) | Cohort 2: Debio 1347 (Urothelial Cancer) (N=4) | Cohort 3: Debio 1347 (All Other Solid Tumor Histologies) (N=29)
Fatigue (General disorders) | 9 | 1 | 10
Pyrexia (General disorders) | 7 | 0 | 1
Oedema peripheral (General disorders) | 4 | 0 | 3
Asthenia (General disorders) | 2 | 0 | 1
Pain (General disorders) | 2 | 0 | 1
Influenza like illness (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 4
Depression (Psychiatric disorders) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 4
Weight decreased (Investigations) | 4 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 3
Platelet count decreased (Investigations) | 3 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 3
Blood bilirubin increased (Investigations) | 2 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 2
Dysgeusia (Nervous system disorders) | 7 | 1 | 9
Dizziness (Nervous system disorders) | 2 | 0 | 2
Headache (Nervous system disorders) | 3 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 9
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0
Dry eye (Eye disorders) | 3 | 1 | 7
Vision blurred (Eye disorders) | 1 | 0 | 3
Lacrimation increased (Eye disorders) | 1 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 0 | 11
Stomatitis (Gastrointestinal disorders) | 9 | 2 | 9
Diarrhoea (Gastrointestinal disorders) | 8 | 0 | 10
Dry mouth (Gastrointestinal disorders) | 11 | 1 | 6
Nausea (Gastrointestinal disorders) | 10 | 0 | 8
Vomiting (Gastrointestinal disorders) | 7 | 1 | 7
Abdominal pain (Gastrointestinal disorders) | 6 | 0 | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 1 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 0 | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 0 | 5
Onychomadesis (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Paronychia (Infections and infestations) | 6 | 0 | 4
Urinary tract infection (Infections and infestations) | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2
Conjunctivitis (Infections and infestations) | 2 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 24 | 2 | 22
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Biliary sepsis (Infections and infestations) | 2 | 0 | 0
Biliary tract infection (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of participants analyzed or technical problems leading to unreliable data.

Due to the premature termination of participant recruitment and shortened follow-up, the primary efficacy analysis was likely underpowered in the final analysis, leading to greater statistical uncertainty in results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or scientific communication related to this study can only take place once the agreement between the Sponsor and the Investigator has been reached.

DOCUMENTS (2):
  • Study Protocol (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03834220/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT03834220/SAP_001.pdf